CLINICAL TRIAL: NCT00436696
Title: Genetic Basis of Neuroblastoma Tumorigenesis
Brief Title: Genetic Analysis Using Blood or Bone Marrow From Participants With Neuroblastoma or Noncancerous Conditions
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL06B1; NCI-2009-00403 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000522985; COG-ANBL06B1; ANBL06B1; ANBL06B1 (Other: Childrens Oncology Group); ANBL06B1 (Other: CTEP)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2017-10

CONDITIONS: Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Recurrent Neuroblastoma; Regional Neuroblastoma; Stage 4 Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, Bone Marrow

GROUPS / COHORTS (1):
- Ancillary-correlative (SNP analysis): DNA samples are derived from participants' banked blood or uninvolved bone marrow. A whole genome scan of DNA samples is employed to identify candidate single nucleotide polymorphisms (SNPs). The candidate SNPs are investigated, using a gene-centric haplotyping approach, to identify 10-20 true disease-associated alleles. The disease-associated alleles are again investigated, using a gene-centric haplotyping approach, to validate 5-10 disease-associated SNPs. SNPs are then analyzed for heritable predisposition.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This laboratory study is looking at genes in participants with neuroblastoma or noncancerous conditions. Identifying genes related to cancer may help in the study of cancer. It may also help doctors predict who is at risk of developing neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Perform a whole genome scan for association of neuroblastoma with single nucleotide polymorphisms (SNP) and SNP haplotypes.

II. Identify true disease-associated SNP alleles using a customized genotyping platform enriched for haplotype analyses in an independent sample set.

III. Validate disease-associated SNP alleles and haplotypes in a final independent sample set.

IV. Identify neuroblastoma predisposition genes.

OUTLINE: This is a multicenter study. Participants are stratified according to presence of high-risk disease (yes vs no) and MYCN amplification (yes vs no).

DNA samples are derived from participants' banked blood or uninvolved bone marrow. A whole genome scan of DNA samples is employed to identify candidate single nucleotide polymorphisms (SNPs). The candidate SNPs are investigated, using a gene-centric haplotyping approach, to identify 10-20 true disease-associated alleles. The disease-associated alleles are again investigated, using a gene-centric haplotyping approach, to validate 5-10 disease-associated SNPs. SNPs are then analyzed for heritable predisposition.

Patients do not receive the results of the genetic testing. A certificate of confidentiality protecting the identity of research participants in this project has been issued by the Children's Oncology Group.

ELIGIBILITY:
Inclusion Criteria:

* Patient:

  * Diagnosis of neuroblastoma

    * Banked constitutional and genomic DNA within COG-ANBL00B1 Neuroblastoma Biology protocol or another COG Biology Protocol
    * At least 1.0 ?g of DNA available
* Control (age, race, and gender-matched):

  * No diagnosis of cancer
  * May have other conditions, including any of the following:

    * Asthma
    * Inflammatory bowel disease
    * Attention-deficit disorder
    * Obesity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 9350 (Estimated)
Dates: Start 2006-12-11 (Actual); Primary Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Neuroblastoma predisposition genes | Up to 4 years
Single nucleotide polymorphism (SNP) allele disease association | Up to 4 years
SNP haplotype disease association | Up to 4 years
Validation of SNP allele and haplotype disease association | Up to 4 years
SNP association with phenotypic subsets (i.e., high-risk vs no high-risk disease; MYCN amplification vs no MYCN amplification) | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: John Maris, Principal Investigator — Children's Oncology Group
Locations (2):
- United States (2):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Childrens Oncology Group, Philadelphia, Pennsylvania